CLINICAL TRIAL: NCT06535412
Title: A Multi-center, Randomized, Double-blind, Placebo Control Phase 1b/II Study to Evaluate the Safety and Efficacy of IMC-002 for the Treatment of Active Systemic Lupus Erythematosus
Brief Title: A Study of IMC-002 for the Treatment of Active Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmuneCare Biopharmaceuticals (Shanghai) Co., Ltd. (Other)
Responsible Party: Sponsor
Organization: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMC002-S-01
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMC-002 + SOC (Experimental)
  Interventions: Drug: IMC-002 + SOC
- Placebo + SOC (Placebo Comparator)
  Interventions: Drug: Placebo + SOC

INTERVENTIONS:
Drug: IMC-002 + SOC — intravenous injection of 0.8mg/kg、1.2mg/kg and1.6mg/kg
  Arms: IMC-002 + SOC
Drug: Placebo + SOC — intravenous injection of Placebo
  Arms: Placebo + SOC

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IMC-002 in the treatment of active SLE.

DETAILED DESCRIPTION:
This is a phase Ib/II study, including 2 stage, phase Ib study to find the dose for phase II study between 0.8mg/kg、1.2mg/kg and 1.6mg/kg dose level, Phase II study is a multi-center, randomized, double-blind, placebo control study to evaluate the safety and efficacy of IMC-002 in active Systemic Lupus Erythematosus patients.

ELIGIBILITY:
Inclusion Criteria:

* Has had a diagnosis of SLE for at least 12 weeks prior to the screening Visit.
* SLEDAI total score ≥ 6 at screening
* BILAG-2004 organ system scores of at least 1 A or 2 B at screening.
* Currently receiving at least one of the SOC SLE medications: oral corticosteroid, antimalarial and/or immunosuppressive agent.
* Other protocol defined inclusion criteria may apply.

Exclusion Criteria:

* Active or unstable neuropsychiatric SLE or lupus nephritis
* Autoimmune or rheumatic disease other than SLE
* Significant, uncontrolled medical conditions not related to SLE
* Active and/or severe viral, bacterial or fungal infection
* History of malignancy within 5 years
* Other protocol defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
SLE Responder Index (SRI-4) | week 52
  Proportion of patients achieving a response in SRI-4

SECONDARY OUTCOMES:
SLE Responder Index (SRI-4) | week 24
  Proportion of patients achieving a response in SRI-4
achieve and sustain a low dose of corticosteroid | week 52
  Proportion of patients who achieve or maintain prednisone </= 7.5 mg/d or equivalent
achieve low level of urine protein | week 52
  Proportion of patients who achieve to reduce urine protein level